# **Carnegie Mellon University**

# **Informed Consent form**

NCT04509024
Incidental Auditory Category Training for Language Learning 1R03HD099382-01

June 5, 2021

#### **Online Consent Form**

**Purpose** This listening task is a research study conducted by Dr. Seth Wiener at Carnegie Mellon University and is funded by Language Learning and the National Institutes of Health. The purpose of the research is to explore new ways to train non-native speakers in a foreign language.

#### **Procedures**

You will be asked to do one of two tasks: 1. identify stimuli presented by a computer and respond on an electronic device or verbally; 2. phonetically transcribe the speech you hear

#### **Participant Requirements**

You must be age 18 or older. For several of our studies, the participant is required to be a Native English speaker, Native Chinese speaker, and/or monolingual, bilingual, dyslexic, right handed, etc. You may be asked about your eligibility below. If you are asked to transcribe speech, you must be able to write in the international phonetic alphabet.

#### Risks & Benefits

The risks and discomfort associated with participation in this study are no greater than those ordinarily encountered in daily life or during routine psychological examinations or tests. Potential risk of breach of confidentiality may occur. There may be no personal benefit from your participation in the study but the knowledge received may be of value to humanity.

### **Compensation & Costs**

The exact amount varies based on length and difficulty of the task. Compensation will not be less than \$1 per hour. A monetary bonus may be included based on the task. There will be no cost to you if you participate in this study.

#### **Confidentiality**

By participating in the study, you understand and agree that Carnegie Mellon may be required to disclose your consent form, data and other personally identifiable information as required by law, regulation, subpoena or court order. Otherwise, your confidentiality will be maintained in the following manner:

Your data and consent form will be kept separate. By participating, you understand and agree that the data and information gathered during this study may be used by Carnegie Mellon and published and/or disclosed by Carnegie Mellon to others outside of Carnegie Mellon. However, any direct personal identifiers will not be mentioned in any such publication of the research data.

Your confidentiality will be maintained during data analysis and publication of results by any or all of the following means: (1) You will be assigned a number as names will not be recorded. (2) The researchers will save the data file by your number, (3) Only members of the research group will view collected data in detail.

## **Carnegie Mellon University**

Note that per regulation all research data must be kept for a minimum of 3 years. This research is being sponsored by the National Institutes of Health, Language Learning, and CMU. These sponsors may access study records.

In the future, once we have removed all identifiable information from your data, we may use the data for our future research studies, or we may distribute the data to other researchers for their research studies. Sharing of data with other researchers will only be done in such a manner that you will not be identified.

Please be aware that any work performed on Amazon MTurk can potentially be linked to information about you on your Amazon public profile page, depending on the settings you have for your Amazon profile. We will not be accessing any personally identifying information about you that you may have put on your Amazon public profile page. We will store your MTurk worker ID separately from the other information you provide to us.

## **Payment Confidentiality.**

Payment methods, especially those facilitated by third party vendors (such as Venmo, Amazon, PayPal), may require that the researchers and/or the vendor may collect and use personal information (first and last name, email addresses, phone numbers, banking information) provided by you in order for your payment to be processed. As with any payment transaction there is the risk of a breach of confidentiality from the third party vendor. All personal information collected by the researcher will be held as strictly confidential and stored in a password-protected digital file, or in a locked file cabinet, until payments are processed and reconciled. This information will be destroyed at the earliest acceptable time.

### **Certificate of Confidentiality**

This research is covered by a Certificate of Confidentiality from the National Institutes of Health. This means that the researchers cannot release or use information, documents, or samples that may identify you in any action or suit unless you say it is okay. They also cannot provide them as evidence unless you have agreed. This protection includes federal, state, or local civil, criminal, administrative, legislative, or other proceedings. An example would be a court subpoena.

There are some important things that you need to know. The Certificate DOES NOT stop reporting that federal, state or local laws require. Some examples are laws that require reporting of child or elder abuse, some communicable diseases, and threats to harm yourself or others. The Certificate CANNOT BE USED to stop a sponsoring United States federal or state government agency from checking records or evaluating programs. The Certificate DOES NOT stop disclosures required by the federal Food and Drug Administration (FDA). The Certificate also DOES NOT prevent your information from being used for other research if allowed by federal regulations.

Researchers may release information about you when you say it is okay. For example, you may give them permission to release information to insurers, medical providers or any other persons not connected with the research. The Certificate of Confidentiality does not stop you from

## **Carnegie Mellon University**

willingly releasing information about your involvement in this research. It also does not prevent you from having access to your own information.

## **Rights**

Your participation is voluntary. You are free to stop your participation at any point. Refusal to participate or withdrawal of your consent or discontinued participation in the study will not result in any penalty or loss of benefits or rights to which you might otherwise be entitled. The Principal Investigator may at his/her discretion remove you from the study for any of a number of reasons. In such an event, you will not suffer any penalty or loss of benefits or rights which you might otherwise be entitled.

## **Right to Ask Questions & Contact Information**

If you have any questions about this study, you should feel free to ask them now. If you have questions later, desire additional information, or wish to withdraw your participation, please contact the Principal Investigator by e-mail:

If you have questions pertaining to your rights as a research participant; or to report objections to this study, you should contact the Research Regulatory Compliance Office at Carnegie Mellon University. Email: <a href="mailto:irb-review@andrew.cmu.edu">irb-review@andrew.cmu.edu</a> . Phone: 412-268-1901 or 412-268-5460.

| You may print a copy of this consent form for your records. |
|---|
| I have no history of hearing impairment. Yes No |
| I am age 18 or older, have read and understand the information above and want to participate. |
| Yes No |